CLINICAL TRIAL: NCT02604745
Title: Degenerative Mitral Regurgitation in Intermediate Risk Patients 65 or Older: Exercise Echocardiogram and HRQOL Post Surgery Preliminary Analysis
Brief Title: Degenerative Mitral Regurgitation in Intermediate Risk Patients
Acronym: DMR
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Principal Investigator, Patrick McCarthy, MD, Chief, Division of Cardiac Surgery, Northwestern University
Other Study IDs: STU00201771
Record Dates: First submitted 2015-11-10; First posted 2015-11-13 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Mitral Valve Insufficiency; Mitral Regurgitation
Keywords: degenerative mitral regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Degenerative Mitral Regurgitation: This cohort includes patients that have had mitral valve surgery for Degenerative Mitral Regurgitation (Type II)

SUMMARY:
The main objective of this project is to determine intermediate-term echocardiographic outcomes in Medicare eligible patients (65 years of age and older) with moderate surgical risk who have undergone mitral valve surgery for degenerative mitral regurgitation.

DETAILED DESCRIPTION:
Severe mitral regurgitation is associated with significant morbidity and mortality. Mitral valve surgical repair has proven to be an effective and durable option in the treatment of symptomatic degenerative mitral regurgitation (MR).

Echocardiography remains a cornerstone in the evaluation of patients with degenerative (Type II) mitral regurgitation allowing for assessment of mitral anatomy, quantification of regurgitant severity, assessment of biventricular function, non-invasive measurement of pulmonary artery systolic pressures and identifying the presence of other valvular disease. The AHA/ACC Valvular Heart Disease Guidelines recommend the use of exercise echocardiography in the setting of mitral regurgitation to determine the degree of mitral regurgitation and pulmonary artery systolic pressures pre and post exercise in addition to an objective determination of the symptoms and exercise capacity.

Echocardiography (both resting and exercise modalities) is helpful in the post-mitral valve repair period in the assessment of the mitral valve gradient and recurrent mitral regurgitation. Symptomatic MR patients can have poor health-related quality of life (HRQOL) which improves and / or returns to comparable age-adjusted norms for reference populations after mitral valve repair or replacement.

To date, there is limited assessment of the degree of mitral regurgitation, mitral stenosis, and exercise capacity following both surgical and percutaneous mitral valve intervention as measured by exercise echocardiography. We propose that this modality with the addition of novel imaging technologies will provide a robust avenue for the assessment of these patients longitudinally. Additionally, assessment of HRQOL, including both the physical and mental health domains, will provide important information with which to guide patient care after mitral valve surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Prior surgery for degenerative mitral regurgitation (DMR) at Northwestern Memorial Hospital performed by a single surgeon.
2. Male and female ≥ 65 years of age at time of index procedure.
3. Mitral Valve surgery performed > 6 months and <36 months at the time of consent. Concomitant procedures at time of index procedure may include incidental CAB, MAZE and tricuspid valve surgery.
4. STS (Society of Thoracic Surgeons) mortality risk score of ≥ 2 and < 6 for mitral valve repair or ≥ 2 and < 8 for mitral valve replacement at time of index procedure.
5. Able to speak, read, and understand English

Exclusion Criteria:

1. Pre-operative tricuspid regurgitation of 4+ (severe) at time of index procedure.
2. Severe RV Dysfunction.
3. Contraindication to exercise testing (i.e., Uncontrolled cardiac arrhythmias causing symptoms or hemodynamic compromise, symptomatic severe aortic stenosis, uncontrolled symptomatic heart failure, etc.).
4. Unable to perform an exercise test due to clinical criteria such oxygen dependency, neuromuscular limitations, NYHA class 4, unstable angina, and postural hypotension.
5. Surgical or interventional cardiac procedure or other intervention since the index procedure that in the opinion of the Investigator may confound data analysis.
6. Left ventricular ejection fraction <30%.
7. Subjects unwilling or unable to give written informed consent.

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with a history of mitral valve surgery for Degenerative Mitral Regurgitation (Type II).
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2021-01 (Actual)

PRIMARY OUTCOMES:
Exercise Capacity | 6 to 36 months Post Index Procedure
  To evaluate exercise duration and workload (METS) in patients who have undergone mitral valve surgery for degenerative mitral regurgitation

SECONDARY OUTCOMES:
Change in HRQOL | Baseline (Index procedure) up to 36 months after surgery
  To determine HRQOL changes from baseline to intermediate term (6 to 36 months) in intermediate risk patients undergoing surgery for Degenerative Mitral Regurgitation
Change in mitral regurgitation | Pre-procedure up to 36 months after surgery
  To determine change in the degree of mitral regurgitation

CONTACTS AND LOCATIONS:
Overall Officials: Patrick M McCarthy, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States